CLINICAL TRIAL: NCT00025220
Title: A Phase II Evaluation of Thalidomide (NSC #66847) in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Thalidomide in Treating Patients With Recurrent or Persistent Cancer of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02415; NCI-2012-02415 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068939; GOG-0231-B (Other: Gynecologic Oncology Group); GOG-0231B (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — Thalidomide

ARMS (1):
- Treatment (thalidomide) (Experimental): Patients receive oral thalidomide once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Thalidomide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Thalidomide — Given PO
  Other Names: THAL
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of thalidomide in treating patients who have recurrent or persistent cancer of the uterus. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor cytostatic activity of thalidomide, as measured by the probability of progression-free survival (PFS) for at least 6 months, in patients with recurrent or persistent uterine leiomyosarcoma.

II. Determine the nature and degree of the toxicity of this drug in these patients.

III. Determine the partial and complete response rates in patients treated with this drug.

IV. Determine the duration of PFS and overall survival of patients treated with this drug.

V. Determine the effect of this drug on initial performance status in these patients.

VI. Determine the effects of this drug at 4 weeks on endogenous angiogenesis factors (vascular endothelial growth factor and basic fibroblast growth factor) in plasma and urine of these patients.

VII. Assess the association of endogenous angiogenesis factors with clinical outcome (PFS) in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary uterine leiomyosarcoma (LMS) that is refractory to curative therapy or established treatments

  * Recurrent or persistent disease
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI OR at least 10 mm by spiral CT scan
  * Tumors within a previously irradiated field are considered non-target lesions
* No smooth muscle tumor of uncertain malignant potential, including metastatic or recurrent disease from such a tumor
* Must have received 1 prior initial chemotherapy regimen (including high-dose, consolidation, or extended therapy after surgical or nonsurgical assessment) for uterine LMS
* Ineligible for a higher priority Gynecological Oncology Group (GOG) protocol (if one exists), including any active phase III protocol for the same patient population
* No documented brain metastases since diagnosis of cancer

  * Patients with stable CNS deficits are allowed provided there are no brain metastases, as confirmed by CT scan or MRI
* Performance status - GOG 0-2 if received 1 prior therapy regimen
* Performance status - GOG 0-1 if received 2 prior therapy regimens
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance greater than 60 mL/min
* No documented seizure disorders since diagnosis of cancer
* Patients with a history of seizure disorders are allowed provided that the seizures have been stable (i.e., no seizure within the past 12 months)while on an appropriately monitored treatment regimen
* No active infection requiring antibiotics
* No greater than grade 1 sensory or motor neuropathy
* No other prior invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant
* Negative pregnancy test
* Fertile patients must use at least 1 highly active method and 1 additional effective method of contraception for at least 4 weeks before, during, and for at least 4 weeks after study participation
* No prior thalidomide
* At least 3 weeks since prior immunologic agents for uterine LMS
* At least 3 weeks since other prior chemotherapy for uterine LMS and recovered
* No more than 1 prior cytotoxic chemotherapy regimen for recurrent or persistent uterine LMS
* No prior non-cytotoxic chemotherapy for recurrent or persistent uterine LMS
* At least 1 week since prior hormonal therapy for uterine LMS
* Concurrent hormone replacement therapy allowed
* At least 3 weeks since prior radiotherapy for uterine LMS and recovered
* No prior radiotherapy to more than 25% of bone marrow
* Recovered from recent prior surgery
* No prior anticancer therapy that would preclude study therapy
* At least 3 weeks since other prior therapy for uterine LMS
* No concurrent bisphosphonates (e.g., zoledronate)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-09; Primary Completion 2003-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
Frequency and severity of adverse effects as assessed by CTC | Up to 7 years

SECONDARY OUTCOMES:
Duration of progression-free survival | Up to 7 years
Duration of overall survival | Up to 7 years
Frequency of clinical response (partial and complete response) | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: D. McMeekin, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States